CLINICAL TRIAL: NCT04731415
Title: Physiologic Change of Posterior Ocular Segment During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HE631577
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Retinal Vascular
Keywords: Retinal vascular density; Optical coherence tomography angiography; Choroidal thickness; Retinal nerve fiber layer thickness; Optic nerve head; Optical coherence tomography
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy pregnant women (Other): Optical coherence tomography and Optical coherence tomography angiography using Optovue® were performed in each trimester and at 6 weeks after childbirth.
  Interventions: Device: Optical coherence tomography and optical coherence tomography angiography (Optovue®)

INTERVENTIONS:
Device: Optical coherence tomography and optical coherence tomography angiography (Optovue®) — Optical coherence tomography and optical coherence tomography angiography (Optovue®) were performed in each trimesters and at 6 weeks after childbirth.
  1. st trimester : gestational age 8-12 weeks
  2. nd trimester : gestational age 24-28 weeks
  3. rd trimester : gestational age 34-38 weeks

SUMMARY:
Women's physiology changes markedly during normal pregnancy. The most distinct alterations occur in the hormonal and cardiovascular systems. There is a dramatic increase in both estrogen and progesterone. Blood volume starts to increase in the first gestational period and reaches a peak in the third trimester.

The physiologic ocular changes during pregnancy are mainly the result of hormonal and blood volume increase, and then are usually marked in the third trimester.

DETAILED DESCRIPTION:
Ocular anterior segment changes during pregnancy are the followings

* Melanogenesis of eyelid and facial skin -> melasma
* Cellular alteration of lacrimal and meibomian gland -> dry eye symptoms
* Increased corneal thickness and corneal curvature -> contact lens intolerance
* Increased lens thickness -> loss of accommodation
* Decreased intraocular pressure -> better glaucoma control There are few studies of posterior changes in pregnant women. Many limitations of previous publications includes lack of internal control and no data of postpartum contraception. However, choroidal thickness seems to be thicker in pregnant women than non-pregnant women. The other changes are non-inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Age > 18 years
* Gestational age < 12 weeks
* Written informed consent

Exclusion Criteria:

* High risk pregnancy such as multifetal pregnancy and preeclampsia
* History of vitreoretinal diseases such as retinal vasculitis
* History of intraocular laser treatments or intraocular surgeries
* History of systemic diseases such as diabetes mellitus and thyroid disease
* Refractive error; spherical equivalence > 4 diopters
* Clear ocular media
* Could not be taken the images by non-dilated pupil

Withdrawal Criteria:

* Preterm labor; gestational age < 34 weeks
* Multifetal pregnancy was demonstrated by ultrasound
* Severe labor and delivery complications such as
* Severe postpartum complications such as postpartum bleeding
* Taking hormone during the follow-up period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Retinal vascular density | 40 weeks
  % of retinal vascular density is measured by optical coherence tomography angiography

SECONDARY OUTCOMES:
Choroidal thickness | 40 weeks
  Choroidal thickness (um) is measured by optical coherence tomography
Retinal nerve fiber layer thickness | 40 weeks
  Retinal nerve fiber layer thickness (um) is measured by optical coherence tomography
Optic disc tomography | 40 weeks
  Cup area and disc area (mm3) are measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No